CLINICAL TRIAL: NCT02562300
Title: Comparative Study of Sublingual Misoprostol Versus Oxytocin in Reducing Bleeding at Cesarean Section
Brief Title: Uterotonics Using to Reduce Bleeding at Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Utrotonics during CS
Record Dates: First submitted 2015-09-27; First posted 2015-09-29 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublingual misoprostol (Active Comparator): The patients in this arm received 400 micrograms of sublingual misoprostol, immediately after delivery of the neonate.
  Interventions: Drug: Misoprostol
- oxytocin (Active Comparator): The patients in this arm received 20 IU oxytocin dissolved in 1 L of Lactated Ringer's or glucose solution) at the rate of 125 ml /h , immediately after delivery of the neonate.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — 400 micrograms of sublingual misoprostol were given immediately after delivery of the neonate.
  Arms: Sublingual misoprostol
Drug: Oxytocin — 20 IU oxytocin dissolved in 1 L of Lactated Ringer's or glucose solution) at the rate of 125 ml /h were given immediately after delivery of the neonate.
  Arms: oxytocin

SUMMARY:
Postpartum haemorrhage continues to be a leading cause of maternal morbidity and mortality worldwide and that is according to the estimates of the World Health Organization in 1998. Average blood loss during delivery progressively increases with the type of delivery, vaginal delivery (500 ml), cesarean section (1000 ml) and emergency hysterectomy (3500 ml) of blood.

A reduction of operative blood loss at cesarean section has a great benefit to the patients in terms of decreased postoperative morbidity and a decrease in risks associated with blood transfusions. The routine use of oxytocin is associated with a significant reduction in the occurrence of postpartum hemorrhage.

Excessive blood loss as estimated by a 10% drop in the hematocrit value postdelivery or by need for blood transfusion, occurs in approximately 4% of vaginal deliveries and 6% of cesarean births.

Although many delivery units use oxytocin as the first line agent to prevent uterine atony at cesarean section, it may not be the ideal agent for prevention of postpartum haemorrhage especially in compromised patients with preeclampsia, cardiac disease or prolonged labor. Oxytocin and specifically its preservative chlorobutanol increases the heart rate and has negative inotropic, antiplatelet and antidiuretic effects.

Misoprostol, a prostaglandin E1 analogue, has been shown in many studies to be an effective myometrial stimulant of the pregnant uterus which binds to prostanoid receptors.

Misoprostol administration, either by oral or rectal route, has been shown to be effective in prevention of postpartum haemorrhage and is considered as an effective alternative to other conventional oxytocics especially in developing countries as it is cheap and thermostable.

Pharmacokinetic studies suggested that the bioavailability of misoprostol after sublingual administration was higher than those after oral or vaginal administration.

A few studies are now available for the use of sublingual misoprostol in the prevention of postpartum haemorrhage following vaginal delivery and have reported it as an effective and convenient route of administration.

However, none of the studies conducted so far have evaluated the response of sublingual misoprostol for prevention of postpartum haemorrhage during cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 37-40 wk.
* Elective lower segment cesarean section.
* Under spinal anesthesia.

Exclusion Criteria:

* Anemia (Hb> 8 g%).
* Multiple gestation.
* Antepartum hemorrhage.
* Poly-hydramnios.
* Two or more previous cesarean sections.
* History of previous rupture uterus.
* Current or previous history of significant disease including heart disease, liver, renal disorders or known coagulopathy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Blood loss in ML | 1 year

SECONDARY OUTCOMES:
Hematocrit value (%) | 1 year